CLINICAL TRIAL: NCT01995747
Title: The Effect of Humanized Anti-CεmX Antibody (h4B12) on IgE Production in the PBMC Isolated From Atopic Dermatitis Patients
Brief Title: The Effect of Anti-CεmX on IgE Production
Acronym: h4B12PBMC
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201109045RC
Record Dates: First submitted 2013-11-21; First posted 2013-11-27 (Estimated); Last update posted 2013-11-27 (Estimated); Status verified 2013-11

CONDITIONS: Atopic Dermatitis
Keywords: IgE; Atopic Dermatitis; antibody; allergy
MeSH Terms: conditions — Dermatitis, Atopic; Hypersensitivity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Despite the success of Omalizumab that neutralizes free IgE in blood and interstitial fluids, treatment of many allergic disorders remains an unmet medical need. Omalizumab was approved for patients having serum IgE levels in the range of 30-700 IU/ml. Omalizumab may not be effective for patients with much higher serum IgE levels, such as those with atopic dermatitis. Therefore, an alternative approach that targets IgE-committed B cells directly and inhibits the synthesis of IgE without binding to free IgE will be attractive. Anti-CεmX mAb, developed by Dr. TW Chang in Academia Sinica, binds human mIgE+ cells, including IgE-committed lymphoblasts and memory B cells. Such anti-CεmX mAbs should be able to activate B cell receptor (BCR) signaling, which leads to anergy or apoptosis of mIgE+ B lymphoblasts, and induces ADCC through their Fc portion. Depletion of mIgE+ B cells by anti-CεmX treatment would inhibit the formation of IgE-producing plasma cells, resulting in a long-term attenuation of IgE synthesis that would eventually lead to a desensitized state in allergic patients.

DETAILED DESCRIPTION:
This study will collect blood from patients of high serum IgE levels to investigate the function of h4b12, a humanized mAb specific for mIgE+ B cells, and compare the effects of h4B12, Omalizumab, and Rituxumab on the suppression of IgE production and the number of IgE-producing plasma cells. These blood specimens will be collected from 50 patients of atopic dermatitis or urticaria with high serum IgE levels. Fountain Biopharma will carry out the following two in vitro assays to measure the efficacy of h4B12:

* IgE ELISA to determine the concentration of IgE.
* IgE ELISPOTto determine the number of IgE-producing plasma cells.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects aged ≥ 18 years
* Clinical diagnosis of atopic dermatitis or chronic urticaria

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients of atopic dermatisis
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2012-02; Primary Completion 2012-06 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
IgE | Day 14
  mesure IgE production in PBMC culture supernatant

CONTACTS AND LOCATIONS:
Overall Officials: Chia-Yu Chu, M.D., Ph.D., Principal Investigator — Dept of Dermatology, NTUH
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan, Taiwan